CLINICAL TRIAL: NCT02692599
Title: A Blind, Randomized and Controlled Clinical Trial With Live Attenuated Mumps Vaccines in Healthy Infants
Brief Title: Safety and Immunogenicity Study of Live Attenuated Mumps Vaccines in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sinovac (Dalian) Vaccine Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-MUMPS-3001
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-04

CONDITIONS: Mumps
Keywords: live attenuated mumps vaccine; safety; immunogenicity; infant
MeSH Terms: conditions — Mumps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): * Single intramuscular injection of the investigational vaccine (0.5 ml) on Day 0;
  * Intervention: investigational live attenuated mumps vaccine;
  Interventions: Biological: investigational live attenuated mumps vaccine
- Control Group (Active Comparator): * Single intramuscular injection of the control vaccine (0.5 ml) on Day 0;
  * Intervention: control live attenuated mumps vaccine;
  Interventions: Biological: control live attenuated mumps vaccine

INTERVENTIONS:
Biological: investigational live attenuated mumps vaccine — The investigational vaccine was manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd.
  Arms: Experimental Group
Biological: control live attenuated mumps vaccine — The control vaccine was manufactured by Zhejiang VACN bio-pharmaceutical Co. Ltd.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of a live attenuated mumps vaccine in healthy infants between 8 - 18 months old with a commercialized live attenuated mumps vaccine as the control vaccine.

DETAILED DESCRIPTION:
This study is a randomized, blind, single-center, controlled phase III clinical trial. The purpose of this study is to evaluate the immunogenicity and safety of a live attenuated mumps vaccine manufactured by Sinovac (Dalian) Vaccine Technology Co., Ltd. The control vaccine is a commercialized live attenuated mumps vaccine manufactured by Zhejiang VACN bio-pharmaceutical Co. Ltd. All participants are healthy infants between 8 - 18 months old, and will be randomly assigned into experimental group or control group in the ratio 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer between 8 - 18 months old;
* Proven legal identity;
* Guardian(s) of the volunteer should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study;
* Complying with the requirement of the study protocol;

Exclusion Criteria:

* Axillaty temperature > 37.0 °C;
* Any significant abnormity of heart, lung, liver, spleen, lymph nodes, or pharynx;
* Acute disease or acute stage of chronic disease within 7 days prior to study entry;
* Prior vaccination with mumps vaccine or with history of mumps infection;
* History of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) about vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc;
* Receipt of any of the following products:

  1. Any subunit vaccine or inactivated vaccine within 14 days prior to study entry;
  2. Any live attenuated vaccine within 28 days prior to study entry;
  3. Any other investigational medicine(s) within 30 days prior to study entry;
  4. Blood product (e.g., immunoglobulin) within 3 months prior to study entry;
  5. Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within 6 month prior to study entry;
* Epilepsy (except febrile seizures), history of seizures or convulsions, or a family history of mental illness;
* Autoimmune disease or immunodeficiency;
* Congenital malformation, developmental disorders, or serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders;
* Severe malnutrition;
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities);
* Any other factor that suggesting the volunteer is unsuitable for this study based on the opinions of investigators;
* Participants with the following conditions between day 0 - 28 of this study would be included in the full analysis set (FAS), but would be excluded from the per protocol set (PPS):

  1. Receipt of any other investigational or unregistered product (drug or vaccine);
  2. Receipt of immunosuppressant (corticosteroid dosage that equivalent to or above 0.5 mg prednisone/kg weight/day) for > 14 days consecutively, except for inhalant or locally administrated corticosteroid;
  3. Receipt of immunoglobulin and/or blood product;
  4. Newly diagnosed autoimmune disease or immunodeficiency (e.g., HIV infection);

Ages: 8 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1150 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of susceptible subjects in each group | 28 days
  Subjects whose pre-immune HI antibody level < 1:2 are considered susceptible; among these subjects, those with post-immune HI antibody level ≥ 1:2 are considered seroconverted.

SECONDARY OUTCOMES:
The incidences of adverse events (AEs) of each group | 28 days
  AEs occurred within 28 days after injection will be collected.
The incidences of serious adverse events (SAEs) of each group | 28 days
  SAEs occurred within 28 days after injection will be collected.
The post-immune geometric mean titers (GMTs) of susceptible subjects in each group | 28 days
  Subjects whose pre-immune HI antibody level < 1:2 are considered susceptible.
The overall SCRs of each group | 28 days
  Subjects whose pre-immune HI antibody level < 1:2 and post-immune antibody level ≥ 1:2, or those whose pre-immune antibody level ≥ 1:2 and the increase of post-immune HI antibody level ≥ 4 folds are considered seroconverted.
The overall post-immune GMTs of each group | 28 days
  The GMTs of all the subjects in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Jingchen Ma, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Dingxing County Center for Disease Control and Prevention, Baoding, Hebei, China

IPD SHARING:
Plan to Share IPD: No